CLINICAL TRIAL: NCT00744601
Title: Impulsivity, Neural Deficits, and Relapse in Cocaine Addiction
Brief Title: Impulsivity, Neural Deficits and Cocaine Addiction
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bryon H Adinoff, Professor, University of Texas Southwestern Medical Center
Other Study IDs: DA023203; 1R01DA023203-01 (NIH)
Record Dates: First submitted 2008-06-19; First posted 2008-09-01 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Cocaine Dependence
Keywords: impulsivity; cocaine dependence; relapse; neuroimaging; functional magnetic resonance imaging (fMRI); single photon emission computed tomography (SPECT)
MeSH Terms: conditions — Cocaine-Related Disorders; Impulsive Behavior; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — urine, blood, plasma, and erythrocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with Cocaine Addiction
- 2: Healthy Control Volunteers

SUMMARY:
The purpose of this study is to assess neurocognitive and associated neural regions/circuitry disruptions relevant to impulsive relapse in cocaine-addicted subjects, and the relationship of the cognitive and neural mechanisms of impulsivity/decision-making to relapse style.

DETAILED DESCRIPTION:
This study is designed to explore putative differences in impulsive behaviors and decision making in cocaine-addicted and healthy control subjects using functional magnetic resonance imaging (fMRI), single photon emission tomography (SPECT), and neurocognitive tasks. We predict that cocaine-addicted subjects will demonstrate neurocognitive and neural alterations in measures of impulsivity and decision-making when compared to healthy controls. That is, cocaine-addicted subjects will show both decreased activation and decreased resting measures of regional cerebral blood flow (rCBF) of the brain structures associated with impulsivity and decision-making. Furthermore, neurocognitive and neural deficits associated with impulsivity and decision-making will be associated with each other and with measures indicative of an impulsive relapse and altered decision making.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine-dependence (patient population) or no cocaine-dependence (control population).

Exclusion Criteria:

* Other medical or psychiatric disorders that may effect neural functioning.
* Medications that may effect neural functioning.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from residential treatment programs at the VA North Texas Health Care System, Nexus Recovery Inc., and Homeward Bound Inc. Healthy controls will be recruited from the Greater Dallas community.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Determine if the brain regions involved in inhibition and decision-making are altered in cocaine-addicted subjects compared to healthy controls. | 2 weeks
In cocaine-addicted subjects, determine if neural deficits during disinhibition or decision-making are related to relapse following treatment. | 6 months

SECONDARY OUTCOMES:
Assess the predictive validity of self-report measures of impulsive relapse. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bryon Adinoff, MD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Divison on Addictions, Dallas, Texas, United States